CLINICAL TRIAL: NCT03574194
Title: Methionine-Restricted Diet to Potentiate The Effects of Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended due to COVID-19 pandemic
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU010518
Record Dates: First submitted 2018-06-15; First posted 2018-06-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Lung Cancer; Prostate Cancer; Breast Cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 6-10 weeks methionine-restricted diet (MRD) with standard of care curative-intent radiation therapy (6 week course or less), without concurrent chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methionine-restricted diet (Experimental): 6-10 weeks methionine-restricted diet (MRD) curative intent radiation therapy course of 6 weeks or less.
  Interventions: Dietary Supplement: Methionine-restricted diet

INTERVENTIONS:
Dietary Supplement: Methionine-restricted diet — The methionine-restricted diet diet (MRD) will begin 2 weeks prior to radiation therapy to deplete methionine stores in the body, continue during radiation, and extend for approximately 2 weeks after the last radiation fraction for a total of 6-10 weeks (depending on duration of radiation course).

SUMMARY:
A diet consisting of a reduced quantity of the essential amino acid methionine sensitizes cancer cells to radiation therapy and reduces metastasis formation and disease progression in mice. However, to date, dietary restriction of methionine has not been tested in combination with radiation therapy in humans as a strategy to improve patient outcomes.

DETAILED DESCRIPTION:
Radiation therapy (RT) is often given concurrently with systemic chemotherapy in order to sensitize the cancer cells to radiation and increase local and regional disease control. However, chemotherapy is often associated with significant toxicity and many patients cannot tolerate it. As such, exploring alternative approaches to radiosensitization that may be more tolerable for patients is important. One innovative strategy that has potential to enhance both the safety and efficacy of SBRT is a methionine-restricted diet (MRD) as an adjunct to radiation therapy. While normal cells can tolerate some degree of methionine deficiency, the vast majority of cancer cells are methionine auxotrophs that require dietary intake of methionine. In the absence of methionine, cancer cells undergo cell cycle arrest and cell death. Preclinical data suggests that consuming a reduced quantity of methionine sensitizes cancer cells to radiation therapy and reduces metastasis formation and disease progression in mice; Phase 1 clinical trials have also demonstrated the safety of the diet with and without concurrent chemotherapy; however, dietary restriction of methionine has not been tested in combination with radiation therapy in humans. This protocol will test our hypothesis that a MRD will be a safe addition to radiation therapy for a variety of human malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over age 18
* Any non-skin cancer malignancy to be treated with standard of care, curative-intent, radiation therapy with an RT course of 6 weeks or less, without concurrently administered cytotoxic chemotherapy. Patients with oligometastatic disease being treated with local consolidative radiation therapy are also eligible. Pathologic confirmation of malignancy is not required if the treating physician(s) agree that this lesion is highly likely to be malignant and the patient elects to forego biopsy.
* The RT plan must achieve standard normal tissue dose-volume constraints.
* Zubrod Performance status 0-2
* Adequate organ and marrow function (leukocytes ≥ 2,000/μL, platelets ≥ 50,000/μL, hemoglobin > 8.0 g/dL, total bilirubin ≤ 3 X ULN, AST(SGOT)/ALT(SPGT) ≤ 3 X ULN, albumin > 2.0 g/dL, calcium < 10.5 mg/dL, creatinine ≤ 3 X ULN)
* Negative serum or urine pregnancy test within 72 hours prior to registration for women of childbearing potential
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control, such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills, throughout their participation in the treatment phase of the study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation therapy that would result in overlap of radiation fields.
* Unintentional weight loss of >10% of normal body weight over a period of 6 months or less.
* Use of an appetite stimulant in the past 6 months for unintentional weight loss.
* Allergy to soy (an ingredient in both methionine-free medical food supplements).
* Administration of cytotoxic chemotherapy within 4 weeks prior to initiation of the study treatment.
* Use of ongoing biologic/targeted/immune/hormonal therapy will be permitted.
* There should be no intention for the patient to receive other local therapy (radiotherapy and/or surgery) or cytotoxic chemotherapy within 4 weeks after completion of the study treatment
* Active systemic, pulmonary, or pericardial infection.
* Psychiatric illness/social situations that would limit compliance with study requirements. * - Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of combined MRD plus RT will be assessed by measuring the rate of 1-year grade 3 or higher adverse events definitely, probably, or possibly related to MRD and RT, using CTCAE version 5.0. | One year from the start of methionine-restricted diet (MRD)
  The expected cumulative rate of grade 3-5 toxicity is less than 15%

SECONDARY OUTCOMES:
Patient adherence to the MRD will be assessed by measuring plasma methionine levels 2 weeks and 6 weeks after starting the MRD | Measurements will be done 2 weeks and 6 weeks after starting the MRD
  Plasma methionine levels less than 13 uM will be considered compliant

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Weir, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Cancer Institute - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-10-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03574194/ICF_000.pdf